CLINICAL TRIAL: NCT01568255
Title: Is Treatment of Vitamin D Deficiency Associated With Resolution of Statin-Induced Muscular Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Margo B. Minissian, Executive Director, Brawerman Nursing Institute, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23187
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Myopathic Symptoms
Keywords: myopathic symptoms
MeSH Terms: interventions — Ergocalciferols

STUDY DESIGN:
Intervention Model Description: The study was prospective, randomized, and double blinded pilot Ergocalciferol 50,000 IU once weekly for 8 weeks compared to Placebo in statin myalgic women. Subjects screened for eligibility underwent baseline and exit visits. For baseline and exit visits, subjects had safety labs drawn for lipid and vitamin D levels, completed Brief Pain Inventory (BPI) severity and interference questionnaires, as well as a Short Form (SF-12) questionnaire and medical history.Additionally, subjects underwent physical exams for baseline visits. After physical exams, subjects were then randomized to Placebo or Ergocalciferol treatment.
Who Masked: Participant, Investigator
Masking Description: This is a randomized, double-blinded, and placebo-controlled pilot study of13 females with moderate to severe myopathic pain while on statins who were enrolled and randomized at a 1:1 ratio.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D Treatment (Experimental): Vitamin D Treatment Group
  Interventions: Drug: Ergocalciferol
- Placebo Group (Placebo Comparator): Placebo at 50,000IU for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergocalciferol — Ergocalciferol therapy at 50,000IU for 8 weeks
  Arms: Vitamin D Treatment
Drug: Placebo — placebo at 50,000IU for 8 weeks
  Arms: Placebo Group

SUMMARY:
Statins are a class of drugs that are highly effective at lowering cholesterol levels. However, compliance is often limited by symptoms of muscle pain. The investigators would like to study Vitamin-D deficient individuals who also have muscle pain due to statin use. About 1 billion people are estimated to have low or insufficient levels of vitamin D worldwide. Patients with low or insufficient levels of vitamin D may develop muscle disease. The purpose of this study is to identify if these symptoms are associated with vitamin D deficiency, and most importantly, if treatment of vitamin D deficiency can reduce muscle pain that is caused by statin treatment.

DETAILED DESCRIPTION:
Vitamin D2 (Ergocalciferol) is approved by the FDA to treat Vitamin D deficiency and will be given according to approved labeling. This drug has not been systematically studied to test the potential benefits of Vitamin D in patients who suffer from statin-induced muscle pain. Vitamin D2 is the current standard of care for treating vitamin D deficiency. Since the investigators are using Vitamin D2 therapy to treat vitamin D deficiency, and because our trial is a pilot study, the data will not be submitted to the FDA for consideration of changing the labeled indications for Vitamin D2 therapy.

This is a randomized, double-blinded, and placebo-controlled pilot study that will only be performed at CSMC. 40 females with moderate to severe myopathic pain while on Simvastatin will be enrolled in this study and will be randomized at a 1:1 ratio. Patients who will be approached are considering an alternative statin medication as part of their clinical care to address their muscle pain.

Participants will be recruited from the investigators' clinic patients. The study will be discussed with a patient during clinical visit by the treating doctor. Interested individuals will be provided with a copy of the consent form to take home for review with friends, family, and other physicians. The patient may then call the study staff to set a study appointment or enroll in the study during the clinical visit. A study investigator will discuss the study with the patient and ask the patient to read through the consent. The investigator will encourage the patient to ask any questions or discuss any concerns she might have.

If the consenting investigator is also the patient's treating doctor, the consenting investigator will request that the study coordinator approach the patient to determine the patient's interest in the study in order to avoid a conflict of interest. The coordinator will explicitly tell the patient that the patient's participation in the study is completely voluntary and that the patient's medical care will not be affected should she choose not to participate.

Participation in this study will be approximately 8 weeks. 20 participants will be randomized to the treatment group and 20 to the placebo group. The treatment group will receive Vitamin D2 therapy at 50,000 IU for 8 weeks (once per week) while the placebo group will receive a placebo pill (once per week) that is identical in nature. Participants have 2 study visits respectively at Week 0 and Week 8, and 1 phone follow-up visit at Week 1. In addition to the administration of Vitamin D2 or placebo mentioned above, other study procedures include informed consent, physical exam, questionnaires (brief pain assessment, and SF-12 to assess limitations on physical activity), review of medical records, medication and supplement review, blood draw, and phone followup. Subjects will be asked to stop any supplemental Vitamin D therapy to maintain an equal dose within patients in the Vitamin D2 and placebo group.

Prior to randomization, statin medication will be changed from Simvastatin to Atorvastatin and patients will be followed up by telephone at Week 1 for tolerability of the new statin medication. When a patient is intolerant to a particular statin, it is the standard of care to attempt another statin medication. Typically, many choose atorvastatin since a lower dose of the drug can be used to obtain the same target LDL/HDL, and lower doses reduce the risk of toxicity. This change in medication would be preformed regardless of the research protocol. Since the statin will be switched to a lower dose, it is possible that it will be a confounding factor, however, even the placebo group will be switched to the same alternate statin, reducing the differences between the two groups. In addition, Atorvastatin is also metabolized by the CYP3A4 enzyme, and because the presumed mechanism of association between vitamin D deficiency and statin-induced myopathic pain pivots on this enzyme, the investigators wanted to choose a statin that continues to utilize this enzyme. But, for reasons stated above, Atorvastatin has less myopathic symptoms due to lower doses used.

At the conclusion of the study, those in the treatment group whose serum 25 OH D levels have reached > 30ng/mL (therapeutic) may continue on maintenance doses on ergocalciferol (1,000 Units/day) if they are receiving clinical benefit. For those whose 25 OH D levels are < 30ng/mL, regardless of whether they received clinical benefit or not from the treatment arm, they will be offered a repeated 8 week course of Ergocalciferol therapy at 50,000 Units/week under standard of care. It will be up to the patient to accept or decline the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender (refer to section 4)
2. Age > 18, using an effective form of contraception (refer to section 4)
3. An indication to be on statin therapy
4. Moderate to severe myopathic pain while on Simvastatin
5. Serum CK level < 10 x ULN
6. Vitamin 25 OH D level < 30 ng/mL (as secondary hyperparathyroidism is triggered below this level)1
7. English speaking patients only
8. Myopathic pain that cannot be attributed to other medical conditions
9. Continue a statin within the CYP3A4 family
10. Competent to give informed consent

Exclusion Criteria:

1. Clinical diagnosis of overt vitamin D deficiency: osteomalacia, rickets, hypocalcemia, hypophosphatemia
2. Already taking Vitamin D supplements > 1000 IU/day
3. Serum creatinine > 2.2 mg/dL within last 6 months
4. AST/ALT > 3 x ULN of the local reference range
5. Serum CK level > 10 x ULN
6. Systolic blood pressure < 100 mmHg
7. Albumin adjusted calcium > 2.55 mmol/L or < 2.20 mmol/L
8. Renal osteodystrophy
9. Malabsorption syndrome
10. Metastatic malignancy
11. Transplant recipients
12. A co-existent diagnosis of renal calculi within the previous 6 months
13. A co-existent diagnosis of primary hyperparathyroidism within the previous 6 months
14. Recent therapy with corticosteroids within the previous 6 months
15. Currently consuming Digoxin, as usage increases risk of hypercalcemia
16. Lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margo B. Minissian, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data was presented by poster presentation internally at Cedars-Sinai Medical Center. The plan is to publish the manuscript.
Supporting Information: Study Protocol, ICF
Time Frame: The data is currently available
Access Criteria: We plan to submit manuscript for peer review.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D Treatment | Placebo Group
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D Treatment | Placebo Group | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11
History of Diabetes [Count of Participants; unit: Participants] — Population: 5/6 placebo participants provided an answer to history of diabetes. 1/6 placebo participants did not provide an answer to history of diabetes
  Participants
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 2 | 2 | 4
History of High Cholesterol [Count of Participants; unit: Participants] — Population: 5/6 placebo participants provided an answer to history of high cholesterol. 1/6 placebo participants did not provide an answer to history of high cholesterol
  Participants
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 4 | 3 | 7
History of High Blood Pressure [Count of Participants; unit: Participants] — Population: 5/6 placebo participants provided an answer to a history of high blood pressure. 1/6 participants did not provide an answer to a history of high blood pressure
  Participants
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 3 | 1 | 4
History of High Triglyceride [Count of Participants; unit: Participants] — Population: 5/6 placebo participants provided an answer to history of high triglycerides. 1/6 placebo participants did not provide an answer to a history of high triglycerides
  Participants
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 2 | 2 | 4
Family History of Coronary Heart Disease [Count of Participants; unit: Participants] — Population: 4/5 Vitamin D participants provided an answer to family history of coronary heart disease. 4/5 Vitamin D participants did not provide an answer to family history of coronary heart disease. 4/6 placebo participants provided an answer to family history of coronary heart disease. 2/6 placebo participants did not provide an answer to family history of coronary heart disease.
  Participants
    number analyzed (Participants) | 4 | 4 | 8
    (all) | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction in Myopathic Pain
Description: To investigate if Vitamin D therapy reduces myopathic pain in subjects on statin medication who have low vitamin D levels and experience myopathic pain.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D Treatment | Placebo Group
Number analyzed (Participants) | 5 | 6
Participants | 4 | 4

2. Primary Outcome: Brief Pain Inventory (BPI) Severity at Exit
Description: Brief Pain Inventory (BPI) severity and interference questionnaires. BPI Severity Scale from 0 (Low Pain) to 10 (High Pain).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D Treatment | Placebo Group
Number analyzed (Participants) | 5 | 6
score on a scale | 4.5625 (2.6877) | 3.8125 (2.4612)

3. Primary Outcome: Vitamin 25 OH D Levels
Description: Assessed with serum measurements
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D Treatment | Placebo Group
Number analyzed (Participants) | 5 | 6
ng/mL | 18.075 (4.537) | 18.05 (6.251)

4. Secondary Outcome: Lipid Profile - Total Cholesterol Levels
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Vitamin D Treatment | Placebo Group
Number analyzed (Participants) | 5 | 6
mg/dl | 165.8 (37.89) | 197.67 (65.68)

5. Primary Outcome: Brief Pain Inventory (BPI) Interference at Exit
Description: Brief Pain Inventory (BPI) severity and interference questionnaires. BPI Severity on a scale from 1 (Low Interference) to 10 (High Interference).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D Treatment | Placebo Group
Number analyzed (Participants) | 5 | 6
score on a scale | 3.85714285725 (1.97948663699) | 0.80952380967 (1.28041234868)

6. Secondary Outcome: Lipid Profile - LDL Cholesterol Levels
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Vitamin D Treatment | Placebo Group
Number analyzed (Participants) | 5 | 6
mg/dl | 88.4 (28.64) | 106.83 (55.33)

7. Secondary Outcome: Lipid Profile - HDL Cholesterol Levels
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Vitamin D Treatment | Placebo Group
Number analyzed (Participants) | 5 | 6
mg/dl | 51.8 (5.72) | 63.5 (18.9)

8. Secondary Outcome: Lipid Profile - Triglycerides Levels
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Vitamin D Treatment | Placebo Group
Number analyzed (Participants) | 5 | 6
mg/dl | 107.54 (0.8943) | 86.92 (128)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Vitamin D Treatment Group: Vitamin D Treatment Group
  Ergocalciferol: Ergocalciferol therapy at 50,000IU for 8 weeks
Arm/Group | Vitamin D Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT01568255/Prot_SAP_000.pdf